CLINICAL TRIAL: NCT04850885
Title: The Co-administration of Dexamethasone or Adrenaline With Lignocaine 2% Prologues Duration in Inferior Alveolar Nerve Block- :A Comparative Study
Brief Title: Efficacy of Dexamethasone or Adrenaline in Inferior Alveolar Nerve Block
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tribhuvan University, Nepal (Other)
Collaborators: National Medical College, Birgunj, Nepal (Unknown)
Responsible Party: Principal Investigator, Dr Saroj Prasad Deo, Associate professor, Tribhuvan University, Nepal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: F-NMC/422/075/076
Record Dates: First submitted 2021-04-12; First posted 2021-04-20 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Oral Surgical Procedure
Keywords: Dexamethasone; Inferior alveolar nerve block

STUDY DESIGN:
Intervention Model Description: The non-probability convenience sampling method was used to select the subjects for this study based on availability and willingness to take part. Total 406 patients presented in department oral and maxillofacial surgery were examined and screened for the study. Detailed history, examination and radiograph ( orthopantomogram) were taken to evaluate disease and mandibular foramina. The sixty subjects were assigned randomly into two groups; DXN or ADN. Subjects were received either Mixture A and Mixture B for IANB on side of surgery. Group ADN has received 4 ml Mixture A ( 2ml Lignocaine 2%+ 2ml freshly prepared solution of adrenaline 0.01mg/ml in normal saline) whereas Group DXN was received 4 ml Mixture B (2ml Lignocaine 2%+ 2ml dexamethasone 4mg/ml).
Who Masked: Participant, Investigator
Masking Description: The blinding of this clinical study was done by confidential supporting staff. The supporting staff was hired for documentation and blinding. Details of role and responsibilities were described to him/her. The study materials ie 30 ml vial of lignocaine 2% (20 mg/ml Xylocaine, AstraZeneca, India); 2 ml in dexamethasone ( 4mg/ml Inj Dexona, Zydus Aliadac, India), in adrenaline 1mg/ml (Actiza, India), normal saline (NS) and identical 5ml syringe and file were given to supporting staff. On the day of surgery, he/she prepared drugs for IANB either the 4 ml Mixture B ( 2ml dexamethasone 4mg/ml + 2ml lignocaine 20mg/ml ) or 4ml Mixture A ( 2ml lignocaine 20mg/ml + 2ml adrenaline 0.01mg/ml, freshly prepared ) in 5 ml identical syringes as mentioned in block randomization chart. The patient name and age were documented the same in a file and a special code was generated and labelled on syringes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone Group ( Group DXN) (Experimental): Group DXN has received 4 ml Mixture B (2ml Lignocaine 2%+ 2ml dexamethasone 4mg/ml)
  Interventions: Drug: inj dexamethasone 4mg/ml and inj lignocaine 20mg/ml
- Adreanaline Group ( Group ADN) (Active Comparator): Group ADN has received 4 ml Mixture A ( 2ml Lignocaine 2%+ 2ml freshly prepared solution of adrenaline 0.01mg/ml in normal saline)
  Interventions: Drug: inj dexamethasone 4mg/ml and inj lignocaine 20mg/ml

INTERVENTIONS:
Drug: inj dexamethasone 4mg/ml and inj lignocaine 20mg/ml — The modified technique of classical IANB was to be selected to avoid failure as described by Clark and Homes (1959). The patients were requested to keep their mouth wide open and an occlusal plane parallel to the floor. Palpation of anatomical landmarks was done properly and the guide finger was positioned at the retromolar fossa. A 5 ml syringe equipped with a 24 gauge needle length of 3.6 cm was used, it was been advanced from premolar on the opposite side into the tissue just above the fingernail until hitting the bone. The body of the syringe was redirected over the lower central incisors and kept parallel to the molars in a horizontal plane at the same time. The needle was inserted another 2 cm deep into the tissue and 3.5 ml of solution X was deposited 1 cm higher than the usual after multiple aspirations (90 degrees two planes). Further, 1 ml solution X was deposited after the withdrawn needle in pterygomandibular space.
  Other Names: inj adreanaline 0.01mg/ml and inj lignocaine 20mg/ml

SUMMARY:
Oral and dental professionals were responsible for the discovery of anaesthesia, given their close day-to-day contact with pain and, hence, their motivation to seek the means to alleviate it. Currently, third molar surgery (TMS) has become the model most frequently used in acute pain trials because third molar surgery (TMS) is simple and frequently used procedure with pain moderate or severe in intensity, as well as sufficient numbers of patients, are available for the required sample size for the studies.

Effective local anaesthesia is arguably the single most important pillar upon which modern dentistry stands. Many agents are not available in the markets of Nepal that provide a rapid onset of surgical anaesthesia with adequate duration. The current study is designed to search for a better quality of perioperative analgesics with a single injection of dexamethasone and lignocaine in IANB preoperatively during TMS. The purpose of the current study is to evaluate the effectiveness and safety profiles of coadministration of dexamethasone (4mg/ml) or adrenaline ( 0.01mg/ml) with lignocaine 2% in IANB during TMS. Best of my knowledge this is a unique and novel clinical trial, probably the first trial which aim to overcome three principal challenges of local anaesthesia with a single injection during TMS.

DETAILED DESCRIPTION:
Background :

Oral and dental professionals were responsible for the discovery of anaesthesia, given their close day-to-day contact with pain and, hence, their motivation to seek the means to alleviate it [Greene NM; 1971]. Currently, third molar surgery (TMS) has become the model most frequently used in acute pain trials because TMS is a simple and frequently used procedure with pain moderate or severe in intensity, as well as sufficient numbers of patients, are available for the required sample size for the studies. Halsted and Hall, 1884 reported the first successful nerve block ie inferior alveolar nerve block and went on to develop nerve and regional blocking techniques [Olch PD, William S; 1975]. These developments in the field of anaesthesia are possibly the most important advances for surgical specialities all over the world. Further, improvements in agents and techniques for local anaesthesia have occurred in the past 100 years. Today's variety of local anaesthetics agents are available can be administered with minimal irritation to tissue but inadequate analgesia, systemic toxicity and adverse local tissue are three principal challenge for clinicians. Local anaesthesia provides benefits of superior pain control, improved patient satisfaction, decreased stress response to surgery, achieve haemostasis, lesser complication with wide therapeutic margins (diminished postoperative nausea and vomiting), decreased logistic requirements, and decrease overall surgical cost. Moreover, clinicians often used local anaesthesia in an effort to improve perioperative analgesia and facilitate early mobilization either as an adjunct to general anaesthesia (GA) or as the primary anaesthetic. LA has become a useful therapeutic approach for managing perioperative pain, ensuring that patients are comfortable enough to be discharged home immediately after third molar surgery, (Robert DH, Sowray JH, 1979).

A broad cross-section of surgical patients consistently ranks postoperative pain as their highest concern highlighting the necessity for prolonged postoperative analgesia [Chew ST. et al, 1998, Razi S. et al 2008]. Usually, analgesia is short-lived, lasting less than 4 hours with all most all local anaesthetic agents. Additionally, the injection technique failure is another challenge to the clinician; past studies were reported the highest failure rate ( 10-39%) with an inferior alveolar nerve block (IANB) [Hung P et al, 2006; Boonsiriseth K et al, 2013]. The researchers have been trying mixing local anaesthetic with adjuvant drugs in an attempt to prolong analgesia from nerve blocks in brachial plexus, femoral, intercostal and interscalene nerve blocks. They found limited success with co-administration of adjuvants such as epinephrine, α2 agonist (i.e. clonidine and dexmedetomidine) opioids, ketamine, midazolam and hyaluronidase [Horliana et al, 2008]. However, co-administration of the dexamethasone was found to be effective for perioperative analgesia in an ample of TMS studies and other nerve blocks study both in the lab and clinical studies.

Effective local anaesthesia is arguably the single most important pillar upon which modern dentistry stands. Many agents are not available in the markets of Nepal that provide a rapid onset of surgical anaesthesia with adequate duration. Local anaesthetic agents that selectively inhibit pain pathways without interrupting transmission of other sensory pathways are not currently available. However, an accident finding of a previous study was impressive to increase the duration of analgesia with lignocaine 2% while the researcher tried to determine the effect of dexamethasone 8 mg on postoperative sequelae after TMS. Following after publication of the result, ample similar studies were conducted and found prolongation in the duration of IANB after injecting dexamethasone in pterygomandibular space. The current study is designed to search for a better quality of perioperative analgesics with a single injection of dexamethasone and lignocaine in IANB preoperatively during TMS. The null hypothesis for this study is "an addition of 2 ml dexamethasone (4mg/ml) or adrenaline ( 0.01mg/ml) to 2ml lignocaine (20 mg/ml) should have same effect of analgesia during TMS''. The purpose of the current study is to evaluate the effectiveness and safety profiles of coadministration of dexamethasone (4mg/ml) or adrenaline ( 0.01mg/ml) with lignocaine 2% in IANB during TMS. Best of my knowledge this is a unique and novel clinical trial, probably the first trial which aim to overcome three principal challenges of local anaesthesia with a single injection during TMS.

Methodology:

Study design:

This study followed Guidelines for Institutional Review Committees (IRCs) for Health Research in Nepal. Approval from the institutional review committee of National Medical College, Birganj of Tribhuwan University, was received before the initiation of this study. To test the study hypothesis, the researcher conducted a prospective, double-blind, randomized, cross-sectional analytical study in a deductive approach. The written informed consent was obtained from all the study participants. The study subject was the American Society of Anesthesiologists (ASA) I-II patients presenting for elective TMS under inferior alveolar block were recruited. The possible risks and benefits of the procedure were described to all the patients. A subject willing for this study was were scheduled for TMS in the morning. Study setting and population:

This quantitative experimental study was conducted in the Department of Oral and Maxillofacial Surgery, National Medical College, Birgunj in between August 2020 to February 2021 and an annual census of approximately 9,000 patients. The sample size calculation was done for comparison between two groups by using the formula; = 2 SD2 (Za/2 +Zβ)2 / d2 where SD [Standard deviation from the previous study], Za/2 [ Standard normal variance to the level of significance (1% type I error, p< 0.01 it is 2.58)], [Zβ = standard normal variance for power ( for 90% power it is 1.28)], d [ effect size ( the difference between the mean value of the previous study) ]. A sample of 27 patients was estimated to give a significant result; however, in this trial were screened 3 times more patient ie 81 patients for the safer side and availability of patient. The patients were enrolled for the study as defined by the sampling criteria. Inclusion criteria were: patients above age 18 who need oral surgery under local anaesthesia and could understand and willing to take part in the study were selected. Non-inclusion criteria were: contraindications to Dexamethasone (i.e., peptic ulcer, renal insufficiency, pregnant women or lactating females ), allergy to NSAIDs ie piroxicam, aged younger than 18 years or older than 85 years, ASA physical status > III, any type of surgery other than a mention, surgery performed under general anaesthesia, patients with any condition precluding the limitation of intra-operative trial drugs ( lignocaine, adrenaline) administration (i.e., significant coronary artery disease, congestive heart failure) or those receiving any premedications (including opioids, benzodiazepines, and clonidine ) or antibiotics or anti-inflammatory drugs within two weeks of the study entry. Also, radiographs showing high and bifid mandibular foramen were non included. Exclusion criteria were: Subject who had to consume analgesic drugs other than the piroxicam 20 mg, whom numbness of tongue and lip was not achieved up to 15 minutes after injection (failure of the block). The subjects did not respond on the VAS scale for 24 hourly and did not come for follow-up for 2nd and 7th postoperatively.

Study Variables:

Predictor variables were: socio-demographic; operative time. Outcome variables were: oedema, trismus, perception of pain in VAS; postoperative analgesia, onset time and duration of anaesthesia. The confounding variables were: stress, the anxiety of subjects, type and degree of difficulty of the operative procedure, the experience of the surgeon. All the surgical procedure were performed by a single experienced surgeon following standard operative protocol which would keep confounding variables fix.

Allocation and randomization of subjects:

The non-probability convenience sampling method was used to select the subjects for this study based on availability and willingness to take part. Total 406 patients presented in department oral and maxillofacial surgery were examined and screened for the study. Detailed history, examination and radiograph ( orthopantomogram) were taken to evaluate disease and mandibular foramina. The sixty subjects were assigned randomly into two groups; DXN or ADN. Subjects were received either Mixture A and Mixture B for IANB on side of surgery. Group ADN has received 4 ml Mixture A ( 2ml Lignocaine 2%+ 2ml freshly prepared solution of adrenaline 0.01mg/ml in normal saline) whereas Group DXN was received 4 ml Mixture B (2ml Lignocaine 2%+ 2ml dexamethasone 4mg/ml). Stratified randomization was done permuted technique of block size 6 and an allocation ratio of 1:1 would lead to random assignment of 3 subjects to Mixture A and 3 to Mixture B. However, subjects were allocated in any of the orders of block after generation of a randomization schedule chart specifying the group to which each subject would be assigned upon the first come first basis. Each block was then randomly chosen to determine the patients' assignment into the groups include all covariates ie age, gender, co-morbidity condition.

Blinding process:

The blinding of this clinical study was done by confidential supporting staff. The supporting staff was hired for documentation and blinding. Details of role and responsibilities were described to him/her. The study materials ie 30 ml vial of lignocaine 2% (20 mg/ml Xylocaine, AstraZeneca, India); 2 ml in dexamethasone ( 4mg/ml Inj Dexona, Zydus Aliadac, India), in adrenaline 1mg/ml (Actiza, India), normal saline (NS) and identical 5ml syringe and file were given to supporting staff. On the day of surgery, he/she prepared drugs for IANB either the 4 ml Mixture B ( 2ml dexamethasone 4mg/ml + 2ml lignocaine 20mg/ml ) or 4ml Mixture A ( 2ml lignocaine 20mg/ml + 2ml adrenaline 0.01mg/ml, freshly prepared ) in 5 ml identical syringes as mentioned in block randomization chart. The patient name and age were documented the same in a file and a special code was generated and labelled on syringes. The investigator ( operator) was received a loaded syringe containing 4 ml clear solution X, either it could be Mixture A or B with special code. The special code was copied to perform while collecting the data. Both surgeon (investigator) and subjects were blinded. The operator used the same syringe contain clear solution X for IANB in the same site of surgery.

Drugs preparation: Freshly prepared mixture of adrenaline or dexamethasone with lignocaine was used in this study for both groups. Preparation of trial drugs for Group ADN, 1 ml solution of in Adrenaline (1mg/ml) was withdrawn in 10 ml syringe and it was diluted to 9 ml of normal saline. From this solution, only 1 ml solution was transferred to a 5 ml syringe and it was diluted to 5ml normal saline. Now, this freshly prepared homogenous mixture of adrenaline (0.02mg/ml). Then 3 ml freshly prepared in adrenaline was discarded from the 5ml syringe and 2ml lignocaine (20mg/ml) was added into the same syringe that was named mixture A. Similarly, mixture B was prepared in an identical 5 ml syringe by withdrawing 2ml lignocaine (20mg/ml) and 2ml of dexamethasone (4mg/ml) that was named as mixture B

Data Collection Technique:

Procedures: The modified technique of classical IANB was to be selected to avoid failure as described by Clark and Homes (1959). The patients were requested to keep their mouth wide open and an occlusal plane parallel to the floor. Palpation of anatomical landmarks was done properly and the guide finger was positioned at the retromolar fossa. A 5 ml syringe equipped with a 24 gauge needle length of 3.6 cm was used, it was been advanced from premolar on the opposite side into the tissue just above the fingernail until hitting the bone. The body of the syringe was redirected over the lower central incisors and kept parallel to the molars in a horizontal plane at the same time. The needle was inserted another 2 cm deep into the tissue and 3.5 ml of solution X was deposited 1 cm higher than the usual after multiple aspirations (90 degrees two planes). Further, 1 ml solution X was deposited after the withdrawn needle in pterygomandibular space. Pre, Intra and post-operative vitals were monitored. Anaesthetic assessment ( subjective and objective) was done as described below. After profound anaesthesia was achieved, a standard surgical procedure for the third molar was performed by the same surgeon. The duration of the operation was recorded as the period between incision given to the last suture placed. Detail of each procedure was recorded. After the surgical procedure, patients were shifted to the postoperative ward for the next 6 hours for observation and further data's collection. Post-operative instructions were given to all patients. They were prescribed Amoxicillin 500 mg (Cap Wymox 500, Pfizer Ltd, India) per oral three times a day for 5 days and piroxicam 20 mg (Fc-tab Dolonex DT, Pfizer Ltd, India) per oral as required as "rescue" analgesia. They were given a sheet of 10 cm visual analogue scale (VAS); (No pain 0-1, Mild pain 2-3, Moderate pain 4-5, Severe pain 6-7, Very severe pain 8-9); were instructed about the rating. They were asked to report to the outpatient setting on the 2nd and 7th postoperative days to observe the surgical outcome and adverse drugs effect on patients. The surgical outcome ie post-facial swelling, trismus and duration of analgesia and drugs adverse reaction ie nausea vomiting, bruise, paraesthesia of lip and tongue, slow wounding, mood change, wound infection, hyperglycemia was recorded these days in our patients' department.

Data Collection Tools: the standard and valid tools were used for the collection of data during the study were the performa and 10 cm visual analogue scale (VAS)(attached in annexe). These tools are reliable and valid and have been increasingly being used to evaluate patients' pain perception.

Assessment:

An armamentarium used for this study were a pulse oximeter (SPO2), thermometer, sphygmomanometer, electric pulp tester, stopwatch. . Supporting staff was given all the above armamentarium and described to prepare test or control group drugs according to the permuted random table. The staff recorded preoperative, intraoperative and postoperative data.

Vital sign and adverse effects assessments:

Pre, Intra and postoperative vitals were recorded with a pulse oximeter (SPO2), non-invasive blood pressure (NIBP) and the respiratory rate which help to assess an adverse effect of drugs. Preoperative and postoperative glucometer random blood sugar (GRBs) was recorded. Wound healing and other local tissue reaction were recorded in 2nd and 7th postoperative days.

Outcome measurements:

A surgical outcome facial swelling (oedema) and trismus were determined by measuring the change in facial contour and inability in mouth opening respectively. Clinical measurements of maximum interincisal distance and facial contours were measured at preoperative day (baseline) and postoperatively days (2nd and 7th day). The facial contour was measured by flexible tape from the tragus to pogonian (Figure ). Similarly, intercessor distance was measured between upper and lower central incisors after asking patients to open the mouth fully with the help of a digital vernier calliper. The examiner was the same one who assessed them preoperatively. Facial oedema and trismus were recorded as the differences between postoperative and preoperative (baseline) values at these appointments.

Postoperative pain is rated on a 10 cm visual analogue scale (VAS) anchored by the verbal description "no pain" (0) and "very severe pain (9)" at every half an hourly up to 24 hours. When the patients began to experience moderate pain (VAS 4-5); it was considered that the anaesthetic effect of the test drugs was terminated. Then patient instructed to take analgesic only prescribed in the researcher. They were asked to record the time every time up to 7 days postoperatively.

Nerve block assessment: IANB was assessed subjectively and objectively. The patients were questioned regarding numbness of lip and tongue a few second after administration of test drugs frequently. Sametime, they were instructed to palpate the lips; compare sensation or numbness in the upper and lower lip. They were asked to report when lower lip numbness had occurred.

The nerve block was assessed objectively every two minute time interval (2, 4, 6, 8, 10 and 15 minute) with an application of cold sprit swabs/ice pack in the lower lip and by the response to atraumatic prick with the blunt instrument in a buccal and lingual mucoperiosteum in relation to 1st molar and canine teeth. The time of complete nerve block was achieved before starting the surgical procedure. The blocks success was standardised that all patients had profound lip numbness. When profound lip numbness was not recorded even after 15 minutes then IANB was considered to be a failure" and such patients were eliminated from the study.

The patients were shifted to the postoperative/ recovery ward adjacent to an ambulatory setting where subjects were observed at least for 6 postoperative hours. The postoperative vitals and ending time numbness and paresthesia of tongue and lip were recorded. The supporting staff rescue the patient with analgesic using in this trial and document the time at which the first analgesic was given after postoperative. Same time, subjects were instructed to palpate the lower lip and tongue every 20 minutes to determine numbness (no feeling) until it returned to normal sensation and asked to note the time. The objective anaesthetic assessment was performed by the investigator at the same time then every hour till the discharge of patients at the 1st molar and canine region. The following data were collected time of local anaesthetic administration; time of analgesia start and lost at 1st molar and canine region; time of lip and tongue numbness start time and regain of sensation started. The duration of IANB was considered the time between the start of operation ie incision to the first analgesic taken. The subjects were instructed not to take any other analgesic drugs and also a total number of analgesics consumes until the 7th postoperative day.

Statistical Analyses:

Data analysis was performed using SPSS statistical software version 11.5 (IBM Corp). The independent Student's t-test analyses were performed for testing hypothesis, groups statistics, comparison between groups. Descriptive analysis was done by calculating frequency and percentages for categorical data. The mean and standard deviation for continuous data. Chi-square test and the Pearson test were applied to determine the association between groups. The confidence level was set at 95%. The significance level was set at < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients above age 18 who need oral surgery under local anaesthesia and could understand and willing to take part in the study were selected.
* contraindications to Dexamethasone (i.e., peptic ulcer, renal insufficiency, pregnant women or lactating females ),
* allergy to NSAIDs ie piroxicam
* ASA physical status > III
* any type of surgery other than a mention surgery performed under general anaesthesia

  --patients with any condition precluding the limitation of intra-operative trial drugs ( lignocaine, adrenaline) administration (i.e., significant coronary artery disease, congestive heart failure)
* those receiving any premedications (including opioids, benzodiazepines, and clonidine )
* antibiotics or anti-inflammatory drugs within two weeks of the study entry. Also, radiograph showing high and bifid mandibular foramen were non included.

Exclusion Criteria:

* Subject who had to consume analgesic drugs other than the piroxicam 20 mg
* The subjects who did not respond on the VAS scale for 24 hourly and did not come for follow-up for 2nd and 7th postoperatively.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
onset time and duration of anaesthesia. | one week post operative
  Postoperative pain is rated on a 10 cm visual analogue scale (VAS) anchored by the verbal description "no pain" (0) and "very severe pain (9)" at every half an hourly up to 24 hours. When the patients began to experience moderate pain (VAS 4-5); it was considered that the anaesthetic effect of the test drugs was terminated. Then patient instructed to take analgesic only prescribed in the researcher. They were asked to record the time every time up to 7 days postoperatively.
  The nerve block was assessed objectively every two minute time interval (2, 4, 6, 8, 10 and 15 minute) with the application of cold sprit swabs/ice pack in the lower lip and by the response to atraumatic prick with the blunt instrument in a buccal and lingual mucoperiosteum in relation to 1st molar and canine teeth. The time of complete nerve block was achieved before starting the surgical procedure. T

SECONDARY OUTCOMES:
post operative facial edema | one week post operative
  A surgical outcome facial swelling (edema) and trismus were determined by measuring change in facial contour and inability in mouth opening respectively. Clinical measurements of maximum interincisal distance and facial contours were measured at preoperative day (baseline) and postoperatively days (2nd and 7th day). The facial contour was measured by flexible tape from the tragus to pogonian (Figure ).
trismus | one week post operative
  Intercessor distance was measured between upper and lower central incisors after asking the patient to open the mouth fully with the help of a digital vernier calliper. The examiner was the same one who assessed them preoperatively. Facial oedema and trismus were recorded as the differences between postoperative and preoperative (baseline) values at these appointments.

CONTACTS AND LOCATIONS:
Overall Officials: Saroj P Deo, 10+2, Principal Investigator — Tribhuvan University, Nepal
Locations (1):
- Saroj Prasad Deo, Birgunj, Two, Nepal

REFERENCES:
- [Background] Deo SP. Effect of submucosal injection of dexamethasone on post-operative sequelae of third molar surgery. JNMA J Nepal Med Assoc. 2011 Apr-Jun;51(182):72-8. PMID 22916516
- [Background] Deo SP. Single-Dose of Submucosal Injection of Dexamethasone Affects the Post Operative Quality of Life After Third Molar Surgery. J Maxillofac Oral Surg. 2016 Sep;15(3):367-375. doi: 10.1007/s12663-015-0846-6. Epub 2015 Dec 7. PMID 27752209
- [Background] Deo SP. Role of addition of dexamethasone to lignocaine 2% with adrenaline in dental nerve blocks for third molar surgery: A prospective randomized control trial. Ann Maxillofac Surg. 2016 Jul-Dec;6(2):260-266. doi: 10.4103/2231-0746.200341. PMID 28299268